CLINICAL TRIAL: NCT00883103
Title: Double Blinded Randomized Trial Between Lidocaine Jelly And Plain Aqueous Gel For Urethral Straight Catheterization And The Q-Tip Test
Brief Title: Double Blinded Randomized Trial Between Lidocaine And Plain Gel For Urethral Straight Catheterization And The Q-Tip Test
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Responsible Party: Oz Harmanli, MD, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 07-091
Record Dates: First submitted 2009-04-15; First posted 2009-04-17 (Estimated); Results first posted 2011-09-13 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-08

CONDITIONS: Pain
Keywords: female urethral catheterization; Lidocaine; lubricant; Q-tip test; Q tip test; K-Y jelly; pain perception; straight catheterization
MeSH Terms: conditions — Pain | interventions — phenylmercury borate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Active Comparator): 2% Lidocaine jelly will be applied onto the catheter and then the cotton swab during evaluation of postvoid residual and the Q-tip test.
  Interventions: Drug: 2% Lidocaine jelly
- Aqueous gel (Placebo Comparator): Plain aqueous gel as placebo will be applied onto the catheter and then the cotton swab during evaluation of postvoid residual and the Q-tip test.
  Interventions: Drug: Plain aqueous gel

INTERVENTIONS:
Drug: 2% Lidocaine jelly — 2% Lidocaine jelly will be applied onto the catheter and then the cotton swab during evaluation of postvoid residual and the Q-tip test.
  Arms: Lidocaine
Drug: Plain aqueous gel — Plain aqueous gel will be applied onto the catheter and then the cotton swab during evaluation of postvoid residual and the Q-tip test.
  Other Names: Surgilube
  Arms: Aqueous gel

SUMMARY:
The purpose of this study is to compare the pain perception between lidocaine and plain aqueous gel during assessment of postvoid residual volume and the Q-tip test.

DETAILED DESCRIPTION:
This study was approved by the institutional review board at Baystate Medical Center. The study pool consists of all women who present to a single urogynecologist's office for an initial consultation with a complaint of urinary incontinence and/or pelvic organ prolapse. Those patients who consent for the research will be then randomized either to 2% Lidocaine Hydrochloride jelly (Akorn, Buffalo Grove, IL) or Surgilube (Fougera, Melville, NY) using computer generated blocks of 10. The latter is a commonly used, commercially available aqueous lubricant gel. Both the urogynecologist who perform the examinations and the patient will be blinded to the randomization. The appearances of the study gels are indistinguishable. Based on our power analysis targeting a power of 0.80, an α value of 0.05, and 20% difference in pain perception between the groups, we are aiming to recruit a sample of minimum132 subjects.

First, demographic information including the age, parity, previous vaginal births, body mass index (BMI), race, diabetes, vaginal atrophy, neurological impairment, current estrogen use, indication for visit and exam anxiety will be collected as a part of patient history. Immediately after voiding, each patient will be placed in a lithotomy position. An independent nurse who is not involved in patient's care will prepare the study gels according to the randomization. After cleansing external urethral meatus with povidone iodine solution, a lubricated a sterile 14-French polyvinyl chloride Mentor Self-Cath catheter (Coloplast, Minneapolis, MN) will be placed transurethrally into the bladder to measure the postvoid residual volume. Following removal of the catheter, a cotton swab, lubricated with the same allocated gel, will be advanced to the urethrovesical junction until resistance was felt. The angle of the Q-tip with the horizontal plane will be measured at rest and with Valsalva maneuver. All the examinations will be performed by the same urogynecologist in the same order. Immediately following the Q-tip test, patient's perception of pain level will be measured using a validated pain scoring system, the Wong-Baker FACES visual scale where 0 represented no pain and 5 represented worst imaginable pain. The rest of the physical examination will be completed after this pain assessment.

We will evaluate patient characteristics and pain score variables by exposure to either Lidocaine or Surgilube using SPSS Version 11.01 software (Chicago, Illinois). For continuous variables, we will calculate the mean and standard deviation and then evaluate significant differences using the Mann Whitney U test. For categorical variables, we will calculate the number and percent and then evaluate significant differences using Pearson's chi-square test. Significance for all results was set at an alpha of <0.05.

ELIGIBILITY:
Inclusion Criteria:

* All women who presented to a single urogynecologist's office for an initial consultation with a complaint of urinary incontinence and/or pelvic organ prolapse

Exclusion Criteria:

* Being a minor
* Pregnancy
* Allergy to Lidocaine or aqueous lubricant gel
* Any current use of analgesia
* Structural abnormalities of the urethra
* Active genital Herpes or other vulvovaginal infections or inability to cooperate with pain assessment due to mental disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oz Harmanli, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

REFERENCES:
- [Result] Harmanli OH, Okafor O, Ayaz R, Knee A. Lidocaine jelly and plain aqueous gel for urethral straight catheterization and the Q-tip test: a randomized controlled trial. Obstet Gynecol. 2009 Sep;114(3):547-550. doi: 10.1097/AOG.0b013e3181b43808. PMID 19701033

RESULTS

PARTICIPANT FLOW:
Groups:
- Lidocaine Gel: 2% Lidocaine jelly will be applied onto the catheter and then the cotton swab during evaluation of postvoid residual and the Q-tip test.
- Placebo: Plain aqueous gel as placebo will be applied onto the catheter and then the cotton swab during evaluation of postvoid residual and the Q-tip test.
Period: Overall Study
Arm/Group | Lidocaine Gel | Placebo
Started | 69 | 68
Completed | 69 | 68
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine Gel | Placebo | Total
Number analyzed (Participants) | 69 | 68 | 137
Age Continuous [Mean (Standard Deviation); unit: years] | 59.9 (12.5) | 57.1 (12.9) | 58.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 68 | 137
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 61 | 62 | 123
  Other | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 69 | 68 | 137
Parity [Mean (Standard Deviation); unit: Previous Live Births] | 2.7 (1.5) | 2.6 (1.5) | 2.7 (1.5)
Previous Vaginal Births [Mean (Standard Deviation); unit: Previous Vaginal Births] | 2.4 (1.6) | 2.4 (1.5) | 2.4 (1.5)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.3 (8.6) | 29.1 (7.8) | 29.2 (8.2)
Diabetes [Number; unit: Participants]
  Yes | 6 | 12 | 18
  No | 63 | 56 | 119
Vaginal Atrophy [Number; unit: Participants]
  Yes | 32 | 31 | 63
  No | 37 | 37 | 74
Neurological Impairment [Number; unit: Participants] — History of stroke, or degenerative vertebral disease without loss of sensation.
  Participants
    Yes | 5 | 6 | 11
    No | 64 | 62 | 126
Current Estrogen Use [Number; unit: participants]
  Yes | 8 | 6 | 14
  No | 61 | 62 | 123
Examination Anxiety [Number; unit: Participants] — Self reported as yes/no by participant, recorded before exam.
  Participants
    Yes | 48 | 48 | 96
    No | 21 | 20 | 41
Indication for the Visit [Number; unit: participants]
  Urinary Incontinence | 35 | 32 | 67
  Pelvic Organ Prolapse | 18 | 22 | 40
  Both | 16 | 13 | 29
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Patient's Perception of Pain Using the Wong-Baker FACES Visual Scale: 0 - no Pain; 5 - Worst Imaginable Pain
Description: A sterile catheter lubricated with the allocated gel was placed transurethrally into the bladder to measure the postvoid residual volume. After removal of the catheter, a cotton swab, coated with the same allocated gel, was advanced to the urethrovesical junction until resistance was felt. The angle of the swab with the horizontal plane was measured at rest and with a Valsalva maneuver. Immediately following the Q-tip test, the patient's perception of pain level was measured by Wong-Baker FACES Pain Scale, a visual scale where 0 represents no pain and 5 represents worst imaginable pain.
Time Frame: Immediately after the examination
Population: All participants assigned to the lidocaine or aqueous gel groups were analyzed. There was no dropout or missing information.
Measure: Median (Full Range); unit: Scores on a scale
Groups:
- Lidocaine: Lidocaine gel was applied to the Q-tip and the catheter before insertion.
- Aqueous Gel: Aqueous gel was applied to the Q-tip and the catheter before insertion.
Arm/Group | Lidocaine | Aqueous Gel
Number analyzed (Participants) | 69 | 68
Scores on a scale | 1 (number) [0 to 5] | 2 [0 to 4]
Statistical Analysis 1: Comparison: Lidocaine vs Aqueous Gel; Test type: Superiority or Other; p < 0.001, Chi-squared

ADVERSE EVENTS:
Arm/Group | Lidocaine Gel | Placebo
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/68
Other Adverse Events (participants affected / at risk) | 0/69 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes